CLINICAL TRIAL: NCT03078101
Title: Effect of Empagliflozin on the Renin-angiotensin System in Patients With Chronic
Brief Title: EMPRA (EMPagliflozin and RAs in Kidney Disease)
Acronym: EMPRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Attoquant Diagnostics (Unknown)
Responsible Party: Principal Investigator, Assoc. Prof. Dr. Manfred Hecking, MD PhD, Assoc. Prof. PD. Dr.med., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EUDRACT-Nr: 2016-002935-14
Record Dates: First submitted 2017-03-07; First posted 2017-03-13 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Diabetic Kidney Disease; Diabetes Mellitus, Type 2; Chronic Kidney Disease stage3; Chronic Kidney Disease stage4
Keywords: Empagliflozin; SGLT-2 Inhibiton and RAS in CKD
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Diabetic CKD patients receiving Empagliflozin 10 MG [Jardiance]
  Interventions: Drug: Empagliflozin 10 MG [Jardiance]
- Group B (Placebo Comparator): Diabetic CKD patients receiving Placebo Oral Tablet
  Interventions: Drug: Placebo Oral Tablet
- Group C (Experimental): Non-diabetic CKD patients receiving Empagliflozin 10 MG [Jardiance]
  Interventions: Drug: Empagliflozin 10 MG [Jardiance]
- Group D (Placebo Comparator): Non-diabetic CKD patients receiving 'Placebo Oral Tablet
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Empagliflozin 10 MG [Jardiance] — administered orally once daily
  Arms: Group A; Group C
Drug: Placebo Oral Tablet — administered orally once daily
  Arms: Group B; Group D

SUMMARY:
This study will be a prospective, clinical pilot study in CKD patients to show whether Empagliflozin in addition to ACEi treatment significantly increases Ang 1-7 levels compared to ACEi treatment alone.

Null and alternative hypotheses:

H0: Empagliflozin in addition to ACEi treatment does not increase Ang 1-7 levels more than ACEi treatment alone.

H1: Empagliflozin in addition to ACEi treatment significantly increases Ang 1-7 levels compared to ACEi treatment alone

Methodology:

Two groups of 24 chronic kidney disease (CKD) patients, respectively, with and without type 2 diabetes will be randomized into the study medication or placebo group. The number of patients per treatment arms is n = 12. Included and consented patients will be subjected to an initial 2-week run-in period for conversion of current RAS blocking medications to ACEi therapy with enalapril or ramipril and respective dose titration to 10 mg enalapril 2 x daily and 10 mg ramipril 1 x daily. Additional antihypertensive medication will be standardized as feasible, with the primary goal of keeping blood pressure as recommended by KDIGO. Following the 2-week run-in phase, all study patients will be subjected to blood collection including the first RAS quantification (RAS Fingerprint) and assessment of HDL composition, as well as urinary analysis and bioimpedance fluid status assessment (BCM measurement). Subsequently, patients will be randomized to either receive empagliflozin (at a dose of 10 mg daily) or placebo. Subsequently, biweekly study visits including electrolyte and glucose (plasma and urine) monitoring as well as BCM measurement will take place. After 12 weeks of study medication intake, a concluding study visit will be scheduled for final RAS quantification (RAS Fingerprint) and HDL analyses as well as final blood and urinary analysis and BCM measurement. Initially, blood and urine will be collected at the clinical visit as part of the routine blood obtainment (no additional effort on patients). From these routine measurements we will be able to extract information regarding the patient's current CKD stage as well as other relevant laboratory parameters (e.g. HbA1c, UACR, etc.). Furthermore, we will document the patient's current medication and significant comorbidities.

Primary analysis variable/endpoint:

The difference of Ang 1-7 increase from baseline between a 3-month treatment with empagliflozin on top of ACEi treatment compared to ACEi treatment alone

Most important secondary analysis variables/endpoints:

1. Simultaneous quantitative changes of multiple RAS effector angiotensin levels determined by mass-spectrometry
2. Recurrence of Ang II levels determined by mass-spectrometry
3. HDL parameters (protein composition of HDL)
4. Renal parameters (albuminuria reduction measured by urinary albumin-creatinine ratio (UACR), renal function (estimated glomerular filtration rate (GFR), serum-creatinine)
5. Urinary electrolyte levels
6. Urinary glucose levels
7. Urinary RAS metabolites (angiotensinogen, ACE and ACE2 levels, ACE2 activity)
8. Blood pressure determined by ambulatory blood pressure measurements
9. Body volume determined by bioimpedance fluid status assessment (BCM measurement)
10. OCR and ECAR in PBMCs determined by Seahorse Flux Analyzer
11. Assessment of reduction of salt sensitivity by using salt sensitivity test with empagliflozin

ELIGIBILITY:
Inclusion Criteria:

for CKD patients with type 2 diabetes

* Estimated GFR (calculated with the MDRD-IDMS formula) between 15 and 59 ml/min (with CKD stage IIIa/b to IV)
* Albumin excretion rates of 30-300 mg/24 hours (UACR <300 mg/g)
* Fasting plasma glucose levels >126 mg/dl [7mmol/L] or HbA1c levels >6.5% (Definition of type 2 diabetes according to the diagnostic criteria set forth by the American Diabetes Association in 2009)

for CKD patients without Diabetes

* Estimated GFR (calculated with the MDRD-IDMS formula) between 15 and 59 ml/min (with CKD stage IIIa/b to IV)
* Albumin excretion rates of 30-300 mg/24 hours (UACR <300 mg/g)

Exclusion Criteria:

CKD patients with type 2 diabetes

* Age <18 years
* Severely impaired renal function (eGFR <15ml/min)
* Hyperkalemia above 4.5mmol/L
* Hypotension (systolic blood pressure lower than 120 mmHg on ambulatory measurement)
* Pregnant patients
* Patients planning pregnancy
* Body mass index < 18.5 kg/m2

for CKD patients without diabetes

* Age <18 years
* Diabetic kidney disease
* Severely impaired renal function (eGFR <15ml/min)
* Hypotension (systolic blood pressure lower than 120 mmHg on ambulatory measurement)
* Pregnant patients
* Patients planning pregnancy
* Body mass index < 18.5 kg/m2 -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
The difference of Ang 1-7 increase from baseline between a 3-month treatment with empagliflozin on top of ACEi treatment compared to ACEi treatment alone | Visit 2 and Visit 8; 3 months
  The difference of Ang 1-7 increase from baseline between a 3-month treatment with empagliflozin on top of ACEi treatment compared to ACEi treatment alone

SECONDARY OUTCOMES:
Mean quantitative changes of baseline multiple RAS effector angiotensin levels after 3 months of empagaliflozin treatment | Visit 2 and Visit 8; 3 months
  Mean quantitative changes of baseline multiple RAS effector angiotensin levels after 3 months of empagaliflozin treatment
Mean changes of baseline Ang II levels after 3 months of empagaliflozin treatment | Visit 2 and Visit 8; : 3 months
  Mean changes of baseline Ang II levels after 3 months of empagaliflozin treatment
Mean changes of baseline specific protein amount on HDL after 3 months of empagaliflozin treatment | Visit 2 and Visit 8; 3 months
  Mean changes of baseline specific protein amount on HDL after 3 months of empagaliflozin treatment
Mean changes in specific renal parameters from baseline in 3 months of empagaliflozin treatment (albuminuria reduction, renal function) | Visit 2 ,3,4,5,6,7,8; 3 months
  Mean changes in specific renal parameters from baseline in 3 months of empagaliflozin treatment (albuminuria reduction, renal function)
Mean changes from baseline relevant blood parameters (HbA1c, β-hydroxybutyrat, elektrolytes, lipids, etc.) after 3 months of empagaliflozin treatment | Visit 2 ,3,4,5,6,7,8; 3 months
  Mean changes from baseline relevant blood parameters (HbA1c, β-hydroxybutyrat, elektrolytes, lipids, etc.) after 3 months of empagaliflozin treatment
Mean changes from baseline urinary RAS metabolites (angiotensinogen, ACE and ACE2 levels, ACE2 activity) after 3 months of empagaliflozin treatment | Visit 2 and Visit 8; 3 months
  Mean changes from baseline urinary RAS metabolites (angiotensinogen, ACE and ACE2 levels, ACE2 activity) after 3 months of empagaliflozin treatment
Mean changes in baseline blood pressure after 3 months of empagaliflozin treatment | Visit 2 ,3,4,5,6,7,8; 3 months
  Mean changes in baseline blood pressure after 3 months of empagaliflozin treatment
Mean changes in body fluid status after 3 months of empagaliflozin treatment | Visit 2 and Visit 8; 3 months
  Mean changes in body fluid status after 3 months of empagaliflozin treatment
Mean changes in baseline oxygen consumption rate (OCR) and the extracellular acidification rate (ECAR) in peripheral peripheral blood mononuclear cells (PBMCs) after 3 months of empagliflozin treatment | Visit 2 and Visit 8; 3 months
  Mean changes in baseline oxygen consumption rate (OCR) and the extracellular acidification rate (ECAR) in peripheral peripheral blood mononuclear cells (PBMCs) after 3 months of empagliflozin treatment
Mean changes in salt sensitivity after 3 months of empagliflozin treatment | Visit 2 and Visit 8; 3 months
  Mean changes in salt sensitivity after 3 months of empagliflozin treatment

OTHER OUTCOMES:
Number of symptomatic hypoglycemia and confirmed hypoglycemic events (plasma glucose level ≤70 mg/dl or an event requiring assistance) | Visit 2 ,3,4,5,6,7,8; timeframe: 3 months
  Number of symptomatic hypoglycemia and confirmed hypoglycemic events (plasma glucose level ≤70 mg/dl or an event requiring assistance)
Number of adverse events reflecting urinary tract infections, genital infections, volume depletion, acute renal failure, bone fractures, diabetic ketoacidosis and thromboembolic events. | Visit 2 ,3,4,5,6,7,8; 3 months
  Number of adverse events reflecting urinary tract infections, genital infections, volume depletion, acute renal failure, bone fractures, diabetic ketoacidosis and thromboembolic events.
Number of cardiovascular events (i.e. stroke, myocardial infarction, heart failure) during the study. | Visit 2 ,3,4,5,6,7,8; 3 months
  Number of cardiovascular events (i.e. stroke, myocardial infarction, heart failure) during the study.
Number of hospitalizations during the study. | Visit 2 ,3,4,5,6,7,8; 3 months
  Number of hospitalizations during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Hecking, MD, Principal Investigator — Department of Internal Medicine III, Division of Nephrology and Dialysis, Medical University of Vienna, Austria
Locations (1):
- Department of Internal Medicine III, Division of Nephrology and Dialysis, Medical University of Vienna, Austria, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818